CLINICAL TRIAL: NCT03005743
Title: COnventional Radiography Based Intracavitary Brachytherapy (Standard Arm) Versus Magnetic Resonance Image Based BrAchyTherapy (Study Arm) in Locally Advanced Cervical Cancers: A Phase III Randomized Controlled Trial (COMBAT - Cervix Trial)
Brief Title: Image Based Brachytherapy in Locally Advanced Cervical Cancers - a Randomized Controlled Trial
Acronym: COMBAT-Cx
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Supriya Sastri (chopra), Professor, Department of Radiation Oncology, ACTREC TATA Memorial Centre Mumbai 410210, Tata Memorial Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMH-1587
Record Dates: First submitted 2016-12-21; First posted 2016-12-29 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; Brachytherapy; Conventional planning; MR based Brachytherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MR based BT (Experimental): Magnetic Resonance Image based Brachytherapy
  Interventions: Radiation: Magnetic Resonance Image based Brachytherapy
- Conventional BT (Other): Conventional Radiograph based Brachytherapy
  Interventions: Radiation: Conventional Radiograph based Brachytherapy

INTERVENTIONS:
Radiation: Magnetic Resonance Image based Brachytherapy — MRI based BT prescription will be in accordance to the GEC-ESTRO guidelines [Intention will be to treat the whole cervix and the remaining residual tumour tissue at the primary site at the time of BT (high risk-clinical target volume) to a dose level analogue to the dose level previously prescribed for point-A]
  Arms: MR based BT
Radiation: Conventional Radiograph based Brachytherapy — The standard conventional radiography based prescription will be according to Manchester system Point A and bladder & rectum ICRU point dose constraints
  Arms: Conventional BT

SUMMARY:
Purpose of the study is to determine whether Image based brachytherapy is superior in terms of local control to Conventional radiograph based brachytherapy in locally advanced cervical cancers in a Phase III randomized setting.

DETAILED DESCRIPTION:
The standard treatment of locally advanced cervical cancer is radio-chemotherapy including external beam radiotherapy (EBRT), brachytherapy (BT) and concomitant chemotherapy with weekly Cisplatin. While image based conformal EBRT is routinely used, prescription and reporting of BT is still based on specific dose points which are conventional radiography based surrogates for tumour (Manchester point A prescription point) and normal tissues [International commission on Radiation Units and Measurements (ICRU) Bladder and Rectum point]. This conventional radiography based planning has been adopted universally for ease of delivering safe doses with reasonably good local control rates (stage IIB - 85%; Stage IIIB - 65%) and acceptable acute and late toxicities (</=10% grade III/IV). Thus, for several decades conventional radiography based prescription has been standard of care universally. But these conventional radiography based surrogates have been proved to be only rough estimates and do not always correlate in 3 dimensional (3D) anatomy for neither tumour nor normal tissues for actual doses delivered and outcomes in terms of control rates and toxicities respectively. Several studies have been published demonstrating limitations and criticizing this point based treatments. In 2006, a working group from Groupe Européen de Curiethérapie- European Society for Therapeutic Radiology and Oncology (GEC-ESTRO) has published recommendations on contouring of tumour target and organs at risk (OAR) as well as on dose volume parameters to be reported for image guided BT in definitive radiotherapy for locally advanced cervical cancer. These recommendations are mainly derived from retrospective single institution experience with Magnetic Resonance (MR) image based Intracavitary Brachytherapy (ICBT). The major advantage of this technique is the possibility to conform the dose given by BT with regard to volume (3D) for both tumour and critical normal tissues (bladder, rectum, sigmoid mainly). Thus, by repetitive imaging performed before each BT treatment it is possible to adapt dose given as per the anatomy of each individual patient taking into account not only the position of OAR but also the tumour regression which often is obtained by preceding EBRT and chemotherapy. Clinical Outcome data from Vienna, Paris and Mumbai have shown potential in improved local control rates with acceptable toxicities so far. Prospectively treated more than 100 patients with image based brachytherapy from Vienna Group have shown improved local control rates across all stages with decreased toxicity on comparisons with historical series of patients treated with Conventional Radiography based BT [13-19]. Also, a phase II multicentre intercontinental study using MR Image Based Brachytherapy (EMBRACE: European study on MRI-guided Brachytherapy in Locally Advanced Cervical Cancer) has been implemented and tested in various centres across the world including Tata Memorial Hospital, Mumbai. Over 600 patients have been recruited in the study so far. Based on the experience collected so far, the image based BT approach is expected to have a major impact on the clinical outcome for II B and III B (increase in local control rates by 10-20%) with concomitant decrease in the rates of late normal tissue toxicity (<5% Grade ¾), as compared to historical results for point based conventional treatment prescriptions [20].

EMBRACE is a study on MRI guided brachytherapy (BT) in locally advanced cervical cancer. Today point-based two-dimensional BT is most often used for definitive radiotherapy in cervical cancer. However, MRI guided Image Based brachytherapy is increasingly being used in several centres, and the results reported so far are very promising. The major advantage of this technique is the possibility to conform the dose given by BT with regard to both volume (3D) and time (4D). Thus, by repetitive imaging performed before each BT implant it is possible to adapt the dose given by BT to the anatomy of each individual patient taking into account not only the position of organs at risk but also the tumour regression which often is obtained by preceding external beam radiotherapy and chemotherapy. Based on the experience collected so far, the image based BT approach significantly improves the dose-volume histogram (DVH) parameters and the improved dose delivered seems to have a major impact on the clinical outcome with a concomitant decrease in the rates of both local failure and morbidity. Preliminary results of ongoing studies including RETRO EMBRACE (600 patients - retrospective multicentric analysis) and EMBRACE (1000 patients recruited so far prospectively multicentric) also suggest excellent local control rates & minimal clinical significant toxicities.

Hypothesis: The clinical outcome of radical radiation therapy including Conventional radiography based brachytherapy for International Federation of Gynecology and Obstetrics (FIGO) Stage IIB and IIIB reported in historical series is 75% and 55% local control rates and grade ¾ rectal / bladder toxicities of 10-15%. With the addition of concomitant cisplatin chemotherapy there is an additional local control benefit of 5-10% and potentially increase in late toxicities (no substantial evidence for toxicities reported so far). With the MR Image Based Brachytherapy approach, mono-institutional series and phase II multicentric international study, the results reported so far show an improvement in local control rates to 96% and 86% for IIB and IIIB respectively and late toxicities <5% reported so far. We propose this randomized control study to test the following hypothesis: With the use of MR Image Based Brachytherapy (Study Arm) in locally advanced cervical cancers (Stratified for Stage IIB and IIIB), there will be an absolute increase in local control rates by 10% and reduction in late rectal and bladder toxicities by 5% - 10% as compared to the Conventional radiography based ICBT. Thus, for demonstrating absolute local control benefit of 10% in Stages IIB (85% to 95%) and Stage IIIB (65% to 75%) a total of 1050 patients (350 patients with Stage IIB and 650 patients with stage IIB respectively) will be accrued.

ELIGIBILITY:
Inclusion Criteria:

* Cancer of the uterine cervix considered suitable for curative treatment with definitive radio-(chemo) therapy including MRI guided Brachytherapy.
* Positive biopsy showing squamous-cell carcinoma, adenocarcinoma or adeno-squamous cell carcinoma of the uterine cervix.
* Stage IIB/IIIB according to FIGO and tumor node metastasis (TNM) guidelines
* Suitable for Brachytherapy boost
* MRI of pelvis at diagnosis is performed
* MRI, Computed Tomography (CT) or Positron Emission Tomography (PET) -CT of the retroperitoneal space and abdomen at diagnosis is performed to rule out Para-aortic lymph node metastasis.
* Patient informed consent
* Pre-treatment Haemoglobin level >10 g/dL

Exclusion Criteria:

* Other primary malignancies except carcinoma in situ of the cervix and basal cell carcinoma of the skin.
* Metastatic disease
* Patients with para-aortic metastatic nodes (stage IVB) to the level of L2 vertebra or further dissemination
* Previous pelvic or abdominal radiotherapy
* Previous total or partial hysterectomy
* Combination of preoperative radiotherapy with surgery
* Patients receiving BT only
* Patients receiving EBRT only
* Patients receiving neoadjuvant chemotherapy
* Contraindications to MRI
* Contraindications to BT
* Active infection or severe medical condition endangering treatment delivery.
* Pregnant, lactating or childbearing potential without adequate contraception

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Local control | 2 years
  Absolute benefit in local control rates by 10% for stages FIGO IIB and IIIB

SECONDARY OUTCOMES:
Late toxicities | 2 years
  Reduction in grade 3 and grade 4 (CTCAE) late toxicities from 10% to 5% (by 50%)
Pelvic control rates | 2 years
Distant failure rates | 2 years
Progression free & cause specific survival | 2 years
Overall survival | 2 years
Quality of life questionnaire EORTC QLQ C30 | 2 years
Quality life questionnaire EORTC QLQ CX24 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Supriya Sastri (Chopra), MD, Principal Investigator — Professor, Department of Radiation Oncology, Tata memorial Hospital, Mumbai 400012
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

REFERENCES:
- [Background] Perez CA, Grigsby PW, Chao KS, Mutch DG, Lockett MA. Tumor size, irradiation dose, and long-term outcome of carcinoma of uterine cervix. Int J Radiat Oncol Biol Phys. 1998 May 1;41(2):307-17. doi: 10.1016/s0360-3016(98)00067-4. PMID 9607346
- [Background] Chemoradiotherapy for Cervical Cancer Meta-analysis Collaboration (CCCMAC). Reducing uncertainties about the effects of chemoradiotherapy for cervical cancer: individual patient data meta-analysis. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD008285. doi: 10.1002/14651858.CD008285. PMID 20091664
- [Background] Vale C, Tierney J, Stewart L. Concomitant chemoradiotherapy for cervical cancer: a systematic review and meta-analysis of individual patient data. Gynecol Oncol. 2006 Feb;100(2):442-3. doi: 10.1016/j.ygyno.2005.09.018. Epub 2005 Oct 17. No abstract available. PMID 16229878
- [Background] Green J, Kirwan J, Tierney J, Vale C, Symonds P, Fresco L, Williams C, Collingwood M. Concomitant chemotherapy and radiation therapy for cancer of the uterine cervix. Cochrane Database Syst Rev. 2005 Jul 20;2005(3):CD002225. doi: 10.1002/14651858.CD002225.pub2. PMID 16034873
- [Background] Kirwan JM, Symonds P, Green JA, Tierney J, Collingwood M, Williams CJ. A systematic review of acute and late toxicity of concomitant chemoradiation for cervical cancer. Radiother Oncol. 2003 Sep;68(3):217-26. doi: 10.1016/s0167-8140(03)00197-x. PMID 13129628
- [Background] Viswanathan AN, Beriwal S, De Los Santos JF, Demanes DJ, Gaffney D, Hansen J, Jones E, Kirisits C, Thomadsen B, Erickson B; American Brachytherapy Society. American Brachytherapy Society consensus guidelines for locally advanced carcinoma of the cervix. Part II: high-dose-rate brachytherapy. Brachytherapy. 2012 Jan-Feb;11(1):47-52. doi: 10.1016/j.brachy.2011.07.002. PMID 22265437
- [Background] Takenaka T, Yoshida K, Tachiiri S, Yamazaki H, Aramoto K, Furuya S, Yoshida M, Ban C, Tanaka E, Honda K. Comparison of dose-volume analysis between standard Manchester plan and magnetic resonance image-based plan of intracavitary brachytherapy for uterine cervical cancer. J Radiat Res. 2012 Sep;53(5):791-7. doi: 10.1093/jrr/rrs033. Epub 2012 Jul 10. PMID 22843369
- [Background] Dolezel M, Odrazka K, Vanasek J, Kohlova T, Kroulik T, Kudelka K, Spitzer D, Mrklovsky M, Tichy M, Zizka J, Jalcova L. MRI-based pre-planning in patients with cervical cancer treated with three-dimensional brachytherapy. Br J Radiol. 2011 Sep;84(1005):850-6. doi: 10.1259/bjr/75446993. PMID 21849368
- [Background] Haie-Meder C, Potter R, Van Limbergen E, Briot E, De Brabandere M, Dimopoulos J, Dumas I, Hellebust TP, Kirisits C, Lang S, Muschitz S, Nevinson J, Nulens A, Petrow P, Wachter-Gerstner N; Gynaecological (GYN) GEC-ESTRO Working Group. Recommendations from Gynaecological (GYN) GEC-ESTRO Working Group (I): concepts and terms in 3D image based 3D treatment planning in cervix cancer brachytherapy with emphasis on MRI assessment of GTV and CTV. Radiother Oncol. 2005 Mar;74(3):235-45. doi: 10.1016/j.radonc.2004.12.015. PMID 15763303
- [Background] Potter R, Haie-Meder C, Van Limbergen E, Barillot I, De Brabandere M, Dimopoulos J, Dumas I, Erickson B, Lang S, Nulens A, Petrow P, Rownd J, Kirisits C; GEC ESTRO Working Group. Recommendations from gynaecological (GYN) GEC ESTRO working group (II): concepts and terms in 3D image-based treatment planning in cervix cancer brachytherapy-3D dose volume parameters and aspects of 3D image-based anatomy, radiation physics, radiobiology. Radiother Oncol. 2006 Jan;78(1):67-77. doi: 10.1016/j.radonc.2005.11.014. Epub 2006 Jan 5. PMID 16403584
- [Background] Potter R, Georg P, Dimopoulos JC, Grimm M, Berger D, Nesvacil N, Georg D, Schmid MP, Reinthaller A, Sturdza A, Kirisits C. Clinical outcome of protocol based image (MRI) guided adaptive brachytherapy combined with 3D conformal radiotherapy with or without chemotherapy in patients with locally advanced cervical cancer. Radiother Oncol. 2011 Jul;100(1):116-23. doi: 10.1016/j.radonc.2011.07.012. Epub 2011 Aug 5. PMID 21821305
- [Background] Mahantshetty U, Swamidas J, Khanna N, Engineer R, Merchant NH, Deshpande DD, Shrivastava S. Reporting and validation of gynaecological Groupe Euopeen de Curietherapie European Society for Therapeutic Radiology and Oncology (ESTRO) brachytherapy recommendations for MR image-based dose volume parameters and clinical outcome with high dose-rate brachytherapy in cervical cancers: a single-institution initial experience. Int J Gynecol Cancer. 2011 Aug;21(6):1110-6. doi: 10.1097/IGC.0b013e31821caa55. PMID 21633296
- [Background] Yoshida K, Yamazaki H, Takenaka T, Kotsuma T, Yoshida M, Furuya S, Tanaka E, Uegaki T, Kuriyama K, Matsumoto H, Yamada S, Ban C. A dose-volume analysis of magnetic resonance imaging-aided high-dose-rate image-based interstitial brachytherapy for uterine cervical cancer. Int J Radiat Oncol Biol Phys. 2010 Jul 1;77(3):765-72. doi: 10.1016/j.ijrobp.2009.05.027. Epub 2009 Oct 14. PMID 19836165
- [Background] Kotsuma T, Yoshida K, Yamazaki H, Takenaka T, Konishi K, Isohashi F, Koizumi M, Tanaka E, Yoshioka Y. Preliminary results of magnetic resonance imaging-aided high-dose-rate interstitial brachytherapy for recurrent uterine carcinoma after curative surgery. J Radiat Res. 2011;52(3):329-34. doi: 10.1269/jrr.10172. Epub 2011 Mar 31. PMID 21467737
- [Background] Beriwal S, Kannan N, Kim H, Houser C, Mogus R, Sukumvanich P, Olawaiye A, Richard S, Kelley JL, Edwards RP, Krivak TC. Three-dimensional high dose rate intracavitary image-guided brachytherapy for the treatment of cervical cancer using a hybrid magnetic resonance imaging/computed tomography approach: feasibility and early results. Clin Oncol (R Coll Radiol). 2011 Dec;23(10):685-90. doi: 10.1016/j.clon.2011.08.007. Epub 2011 Sep 9. PMID 21908180
- [Background] Mahantshetty U, Swamidas J, Khanna N, Engineer R, Merchant NH, Shrivastava S. Magnetic resonance image-based dose volume parameters and clinical outcome with high dose rate brachytherapy in cervical cancers--a validation of GYN GEC-ESTRO brachytherapy recommendations. Clin Oncol (R Coll Radiol). 2011 Jun;23(5):376-7. doi: 10.1016/j.clon.2011.02.006. Epub 2011 Mar 5. No abstract available. PMID 21377847
- [Background] Haie-Meder C, Chargari C, Rey A, Dumas I, Morice P, Magne N. MRI-based low dose-rate brachytherapy experience in locally advanced cervical cancer patients initially treated by concomitant chemoradiotherapy. Radiother Oncol. 2010 Aug;96(2):161-5. doi: 10.1016/j.radonc.2010.04.015. PMID 20655120
- [Background] Schmid MP, Kirisits C, Nesvacil N, Dimopoulos JC, Berger D, Potter R. Local recurrences in cervical cancer patients in the setting of image-guided brachytherapy: a comparison of spatial dose distribution within a matched-pair analysis. Radiother Oncol. 2011 Sep;100(3):468-72. doi: 10.1016/j.radonc.2011.08.014. Epub 2011 Sep 14. PMID 21924510
- [Background] Fidarova EF, Berger D, Schussler S, Dimopoulos J, Kirisits C, Georg P, Bachtiary B, Potter R. Dose volume parameter D2cc does not correlate with vaginal side effects in individual patients with cervical cancer treated within a defined treatment protocol with very high brachytherapy doses. Radiother Oncol. 2010 Oct;97(1):76-9. doi: 10.1016/j.radonc.2010.05.005. Epub 2010 Jun 17. PMID 20561694
- [Background] Sturdza A, Potter R, Fokdal LU, Haie-Meder C, Tan LT, Mazeron R, Petric P, Segedin B, Jurgenliemk-Schulz IM, Nomden C, Gillham C, McArdle O, Van Limbergen E, Janssen H, Hoskin P, Lowe G, Tharavichitkul E, Villafranca E, Mahantshetty U, Georg P, Kirchheiner K, Kirisits C, Tanderup K, Lindegaard JC. Image guided brachytherapy in locally advanced cervical cancer: Improved pelvic control and survival in RetroEMBRACE, a multicenter cohort study. Radiother Oncol. 2016 Sep;120(3):428-433. doi: 10.1016/j.radonc.2016.03.011. Epub 2016 Apr 29. PMID 27134181
- [Background] Prescribing, Recording, and Reporting Brachytherapy for Cancer of the Cervix. J ICRU. 2013 Apr;13(1-2):NP. doi: 10.1093/jicru/ndw027. No abstract available. PMID 27335496